CLINICAL TRIAL: NCT00858013
Title: Multi-center, Randomized, Open Label Study of the Durability of Glycemic Control With Nateglinide Versus Glimepiride as Monotherapy in Type 2 Diabetic Patients
Brief Title: Study of the Durability of Glycemic Control With Nateglinide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Collaborators: Korea University Guro Hospital (Other); Hanyang University (Other); Inha University Hospital (Other); Kyunghee University Medical Center (Other); Myongji Hospital (Other); Bundang CHA Hospital (Other); Wonju Severance Christian Hospital (Other); Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, Kwan Woo Lee, Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AJIRB-CRO-08-197
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Nateglinide; Pancreatic beta cell function
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Nateglinide; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nateglinide (Active Comparator): Nateglinide 90~120mg three times a day
  Interventions: Drug: Nateglinide
- Glimepiride (Active Comparator): Glimepiride 1~2mg once a day
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Nateglinide — Nateglinide 90~120mg three times a day
  Other Names: fastic
  Arms: Nateglinide
Drug: Glimepiride — Glimepiride 1~2mg once a day
  Other Names: amaryl
  Arms: Glimepiride

SUMMARY:
This multi-center, randomized controlled study aims to evaluate the durability and efficacy of nateglinide therapy for long term glycemic control compared with glimepiride.

DETAILED DESCRIPTION:
Selected patients will be randomly assigned to receive nateglinide or glimepiride.

Previous treatment with oral antidiabetic drugs (metformin, a-glucosidase inhibitor, nateglinide or sulfonylurea) will be discontinued. After a 1 month wash-out period (if 6.5 ≤ HbA1c ≤ 8.5), patients will take randomly assigned drugs for 24 months.

Patients will be met by the trial investigator every 3 months following randomization. At each visit, patients whose HbA1c is > 8.0% will be retested 2 weeks later, and if the retested HbA1c is also above 8.0%, those patients will be withdrawn considering monotherapy failure. We will evaluate the durability of nateglinide in comparison with that of glimepiride based on the withdrawal rate.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus
* age>=18years
* no anti hyperglycemic agent for 3 months or low-dose oral hypoglycemic therapy

  * metformin≤1g/day, acarbose≤300mg/day, voglibose≤0.9mg/day, nateglinide≤270mg/day, gliclazide≤80mg/day, glimepiride≤2mg/day, glibenclamide≤5mg/day (nateglinide or sulfonylurea <6months)
* 6.5% ≤ HbA1c ≤ 8.5%

  * patients on no anti hyperglycemic agent for 3 months : HbA1c at screening
  * patients on oral hypoglycemic therapy in 3months : HbA1c after wash-out

Exclusion Criteria:

* attending other clinical trials in 3months
* type I diabetes mellitus
* taking systemic steroid in 1month or requiring steroid therapy during clinical trial
* acute myocardial infarction in 6months
* alcoholics, pituitary or adrenal insufficiency, severe ketosis, diabetic ketoacidosis
* severe liver disease or AST, ALT ≥ 2.5 x ULN
* renal insufficiency (serum creatinine > 2.0mg/dl)
* other severe diabetic complication
* drug hypersensitivity history to nateglinide or sulfonylurea
* pregnant or plan to become pregnant during the clinical trial, lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2009-04-24 (Actual); Primary Completion 2014-06-25 (Actual); Study Completion 2014-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kwan Woo Lee, MD,PhD, Principal Investigator — Ajou University School of Medicine
Locations (7):
- South Korea (7):
  - Hanyang University Medical Center, Guri-si, Gyeonggi-do
  - Myongji Hospital, Ilsan, Kyounggi
  - Inha University Hospital, Incheon
  - Hallym University Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung hee University Medical Center, Seoul
  - Ajou University Hospital, Suwon

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nateglinide | Glimepiride
Started | 46 | 42
Completed | 24 | 23
Not Completed | 22 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nateglinide | Glimepiride | Total
Number analyzed (Participants) | 46 | 42 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (10.5) | 55.1 (12.3) | 55 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 18 | 41
  Male | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: The Durability of Nateglinide in Comparison With Those of Glimepiride Based on the Withdrawal Rate
Description: % monotherapy failure, that means % number of participants who withdrew from the study due to high HbA1c (>8.0%)
Time Frame: every 3 months following randomization, for 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nateglinide | Glimepiride
Number analyzed (Participants) | 24 | 23
Participants | 10 | 7

2. Secondary Outcome: HbA1c
Description: HbA1c (%) at 24 months
Time Frame: at 24 months
Population: data of participants who finished 24 months of follow-up
Measure: Mean (Standard Deviation); unit: % HbA1c
Arm/Group | Nateglinide | Glimepiride
Number analyzed (Participants) | 14 | 16
% HbA1c | 6.9 (0.6) | 6.5 (0.5)

3. Secondary Outcome: Fasting Glucose
Description: fasting glucose (mg/dL) at 24 months
Time Frame: at 24 months
Population: data of participants who finished 24 months of follow-up
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Nateglinide | Glimepiride
Number analyzed (Participants) | 14 | 16
mg/dL | 131.2 (25.9) | 115.7 (19.8)

4. Secondary Outcome: C-peptide
Description: c-peptide(uU/mL) at 24 months
Time Frame: at 24 months
Population: data of participants who finished 24 months of follow-up
Measure: Mean (Standard Deviation); unit: uU/mL
Arm/Group | Nateglinide | Glimepiride
Number analyzed (Participants) | 14 | 16
uU/mL | 1.29 (0.41) | 1.77 (0.72)

5. Secondary Outcome: HOMA-IR
Description: insulin resistance marker HOMA-IR at 24 months
Time Frame: at 24 months
Population: data of participants who finished 24 months of follow-up
Measure: Mean (Standard Deviation); unit: mg/dL x mIU/L
Arm/Group | Nateglinide | Glimepiride
Number analyzed (Participants) | 14 | 16
mg/dL x mIU/L | 2.40 (1.36) | 2.31 (1.70)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Nateglinide | Glimepiride
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 6/24 | 1/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nateglinide (N=24) | Glimepiride (N=23)
hypoglycemia (Endocrine disorders) | 1 | 0
dyspepsia (Gastrointestinal disorders) | 2 | 0
gall stone (Gastrointestinal disorders) | 1 | 0
herpes zoster (Skin and subcutaneous tissue disorders) | 1 | 0
gastritis (Gastrointestinal disorders) | 1 | 0
dizziness (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No